CLINICAL TRIAL: NCT01523548
Title: Carbon Monoxide Therapy for Severe Pulmonary Arterial Hypertension
Acronym: CO in PAH
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding and subject acuity
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Roberto Machado, M.D., Associate Professor of Pulmonary Medicine, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-06425; K23HL098454 (NIH)
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-04

CONDITIONS: Hypertension, Pulmonary
Keywords: Carbon Monoxide; Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Carbon Monoxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carbon Monoxide (Experimental): Inhaled Carbon Monoxide therapy administered over 16 weeks
  Interventions: Drug: Carbon Monoxide

INTERVENTIONS:
Drug: Carbon Monoxide — 150 ppm x 3 hours once weekly (week 1) 150 ppm x 3 hours twice weekly (week 2) 150 ppm x 3 hours three times a week (week 3-16)

SUMMARY:
The purpose of this study is to examine the potential of carbon monoxide (CO) to decrease elevated blood pressure in the pulmonary artery. This symptom is seen in patients with pulmonary arterial hypertension, a rare disease that causes fatigue, dizziness, and shortness of breath because the blood vessels that supply the lungs narrow, forcing the heart to work harder to push blood through. Previous studies in the laboratory have shown that carbon monoxide has promise in treating these symptoms.

Subjects in this study are being asked to undergo a new type of treatment to improve pulmonary arterial hypertension by breathing CO gas. CO is a colorless, tasteless, odorless gas usually found in car exhaust or cigarette smoke. It is administered with a continuous flow of air. Subjects will undergo a screening process during which it will be determined if they are eligible for the study. After the screening process, if subjects meet eligibility criteria for the study, they will begin carbon monoxide treatment through a cushioned mask that is placed over the nose and mouth. This treatment will last for sixteen weeks.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) remains an uncommon debilitating and fatal disease, and is clinically marked by a progressive increase in pulmonary vascular resistance leading to right heart failure and ultimately death. Currently the treatment options available for those suffering from PAH target cellular dysfunction that leads to constriction of the vasculature. Although there is some evidence that available therapies have secondary effects on vascular remodeling there are currently no therapies that target abnormal cell proliferation in PAH.

Carbon monoxide (CO) is a gaseous molecule with known toxicity and lethality to living organisms when exposed to high concentrations for sustained periods. However, CO has shown promise in preclinical models of pulmonary hypertension. Recent studies have shown that mammalian cells have the ability to generate endogenous CO primarily through the catalysis of heme by the heme oxygenase enzymatic system and there is ample evidence demonstrating that CO behaves as a signaling molecule in cellular and biological processes. Furthermore, CO has been demonstrated to exert key physiological and protective functions in various models of tissue inflammation and injury.

This study will evaluate the safety and potential efficacy of inhaled CO in subjects with severe PAH. Over forty subjects with severe PAH despite best available therapy will be screened from the UIC pulmonary vascular disease clinic, of which twenty subjects will be recruited for participation in the trial. The trial will consist of an initial screening period to determine subjects' eligibility for the study. This will be based on a previous echocardiogram, a six minute walk test and right heart catheterization done as part of standard care for subjects with pulmonary arterial hypertension. Following the initial screening, the trial will last sixteen weeks, during which subjects will receive inhaled carbon monoxide up to three times weekly at the University of Illinois at Chicago.

ELIGIBILITY:
Inclusion Criteria:

* male and female ≥ 18 years old , with Pulmonary Arterial Hypertension
* Right heart catheterization diagnosis of PAH:

  * Mean Pulmonary Artery Pressure (mPAP)> 25 mmHg at rest
  * Pulmonary Capillary Occlusion Pressure (PCOP) or Left Ventricular End Diastolic Pressure (LVEDP) < 15 mmHg
  * Pulmonary Vascular Resistance (PVR) > 3 mmHg/L/min
* Must be Class 1.1, 1.2, or 1.3 PAH (see Appendix A)
* Echocardiographic evidence of Right Ventricular Dysfunction
* On standard and stable PAH therapy (no dose changes in the 4 weeks prior to starting the study medication) including:

  * A Prostacyclin (IV epoprostenol, IV or subcutaneous remodulin, inhaled iloprost or remodulin) unless willing or unable to tolerate therapy AND
  * Phosphodiesterase type 5 inhibitor OR
  * Endothelin Receptor Antagonist OR
  * Any combination of a-c
* NYHA class III or IV despite 3 months of stable therapy as outlined above
* 6 minute walk distance ≤ 380m
* Negative serum pregnancy test
* Female of childbearing age either surgically sterilized or using acceptable method of contraception. Acceptable methods of contraception include oral contraceptives, IUD, or other barrier methods of contraception.

Exclusion Criteria:

* History of malignancy in 2 years prior to enrollment
* Baseline cytopenia's:

  * White blood cell count ≤ 3,000 i. Absolute Neutrophil Count (ANC) less than 1500 cells/mm3
  * Hemoglobin ≤ 7
  * Platelet ≤ 100,000
* Baseline Liver Disease:

  * ALT/AST, ALk phos > 2.5x ULN, INR > 1.5
  * Bilirubin > 1.5 x ULN
* Coronary artery disease
* Any cause of pulmonary hypertension other than class 1.1, 1.2, or 1.3 PAH.
* Baseline Renal Disease: Cr ≥ 2
* Active Smoker
* Hypoxemia with SaO2 < 95% on oxygen 2 L/min
* Baseline COHb > 2%
* Pregnancy or lactation
* Inability to attend scheduled clinic visits
* Previous lung transplant
* Naive to available standard PAH therapy
* Pulmonary Capillary Occlusion Pressure (PCOP) or LEft Ventricular End Diastolic Pressure (LVEDP)< 15 mmHg
* Concomitant enrollment in another investigational treatment protocol for PAH or taking any off label drug therapy for PAH
* Recent enrollment in or plans to enroll in Pulmonary Rehabilitation during the study period
* Any condition that in the opinion of the investigator would prevent completion of study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Evidence of a 20% decrease in pulmonary vascular resistance post-therapy when compared to pre-therapy value | At baseline and after 16 weeks

SECONDARY OUTCOMES:
Effect of 16-weeks CO inhalation on other pulmonary and systemic hemodynamic parameters | 16 weeks
Effect of 16-weeks CO inhalation on functional capacity assessed by six-minute walk test | 16 weeks
Effect of 16-weeks CO inhalation on Brain Natriuretic Peptide levels | 16 weeks
Effect of 16-weeks CO inhalation on right ventricular echocardiographic parameters | 16 weeks
Effect of 16-weeks CO inhalation on acute pulmonary vasoreactivity | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roberto F Machado, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago Medical Center, Chicago, Illinois, United States